CLINICAL TRIAL: NCT00599183
Title: Diffusion Tensor (Magnetic Resonance) Imaging and Tractography in Herniation of the Cervical Spine: An Investigator-Initiated Pilot Study
Brief Title: Diffusion Tensor (Magnetic Resonance) Imaging and Tractography in Herniation of the Cervical Spine
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Responsible Party: Principal Investigator, Franklin G. Moser, M.D., Director, Neuro-Interventional Imaging; Vice Chair Radiology Research, Cedars-Sinai Medical Center
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: CSMC IRB PRO00009246
Record Dates: First submitted 2008-01-11; First posted 2008-01-23 (Estimated); Last update posted 2013-07-31 (Estimated); Status verified 2013-07

CONDITIONS: Cervical Spine Herniation
Keywords: Cervical spine herniation; MRI cervical spine; Diffusion tensor imaging cervical spine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Other): Participants will receive baseline conventional MRI of the cervical spine as part of their clinical care with an additional diffusion tensor imaging (DTI)sequence as part of the research; they will complete an anonymized questionnaire about their condition. Participants will receive an MRI with DTI and tractography as part of the research and will complete an anonymized questionnaire about their condition. The baseline and follow up data will be compared.
  Interventions: Other: MRI-Diffusion Tensor Imaging and Tractrography

INTERVENTIONS:
Other: MRI-Diffusion Tensor Imaging and Tractrography — MRI scan: Baseline: Conventional MRI (as part of clinical care) with additional diffusion tensor imaging (DTI)sequence (research). 6-week follow up: MRI with DTI and tractography as part of the research

SUMMARY:
This is an investigator-iniated pilot study to determine if MRI with diffusion tensor imaging (DTI) and tractography will yield useful information in patients suspected of having cervical spine disc herniation to provide imaging confirmation of whether or not disease is progressing and to assess response to treatment (regardless of treatment provided).

DETAILED DESCRIPTION:
Conventional MRI (magnetic resonance imaging) is used to confirm disc herniation of the cervical spine. Symptoms of the condition can change before they can be seen by conventional MR images. Therefore, very little gross change can be seen by conventional MRI even after 6 weeks of treatment, either medical or surgical. This study will investigate whether newer MRI techniques, diffusion tensor imaging (DTI) and tractography, are useful in demonstrating gross changes or assessing response to treatment.

Consenting patients referred for clinically indicated cervical spine MRI by their treating physicians to confirm cervical disc herniation will receive an additional MRI sequence, diffusion tensor imaging. This will provide a baseline. The DTI sequence will add five minutes to the procedure. Participants will return at 6 weeks for a follow up MRI of the cervical spine to include DTI and tractography. Participants will be asked to complete an anonymized questionnaire at enrollment and at follow up to provide information regarding their condition.

MRI is a non-invasive diagnostic study of minimal risk which uses magnets instead of ionizing radiation to acquire images. The images are then assembled by computer. Diffusion tensor imaging (DTI) uses water diffusion to visualize structures in the brain and nervous system. Tractography is performed using DTI and computer post-processing to track the fiber bundles which exist in the brain and spinal cord and visualize them as two and three dimensional images. Both techniques allow radiologists to detect abnormalities, in this case, cervical spine disc herniation.

The follow up studies will be compared to the baseline studies to determine which demonstrates the highest sensitivity and specificity in identifying cervical spine abnormalities in general and cervical spine herniation in particular.

ELIGIBILITY:
Inclusion Criteria:

* Patients suspected of having cervical spine herniation.

Exclusion Criteria:

* Patients not suspected of having cervical spine herniation.
* Patients in which MRI is contraindicated (patients with embedded metallic objects, including pacemakers, surgical clips, spinal cord stimulators, or prosthetic heart valves.)
* Patients requiring general anesthesia or conscious sedation--sedation would increase risk to participants.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2006-08; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Whether DTI alone or with tractography demonstrates greater sensitivity and specificity as a diagnostic tool for this disorder | 6 week follow up scans

CONTACTS AND LOCATIONS:
Overall Officials: Franklin Moser, MD, Principal Investigator — Cedars-Sinai Medical Center
Locations (1):
- Cedars-Sinai Medical Center - S. Mark Taper Foundation Imaging Center, Los Angeles, California, United States